CLINICAL TRIAL: NCT06595810
Title: Exercise Habits and Preferences of Community Dwelling Older Adults with Chronic Pain: an Exploratory Study
Brief Title: Exercise Habits and Preferences of Community Dwelling Older Adults with Chronic Pain
Status: Not yet recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Other Study IDs: EHPP
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Older adult participants: The data collection procedure for the study outlined in the document involves a cross-sectional exploratory approach. The researchers will recruit 20 participants from Neighborhood Elderly Centers and support groups. These participants, who are community-dwelling older adults with chronic pain, will be interviewed individually or in groups. During the 20-minute interviews, they will be asked about their pain situations, including pain intensity and sites of pain, as well as their exercise habits and preferences.

SUMMARY:
Objective:

* To explore the exercise habits and preferences of community dwelling older adults with chronic pain
* To explore the facilitating factors and barriers in performing regular exercise for community dwelling older adults with chronic pain

Significance of study:

Chronic pain is a significant issue affecting both physical well-being and socioeconomic aspects across different age groups. Among older adults, physical inactivity is common, especially among those experiencing chronic pain. However, regular physical exercise offers numerous health benefits for the musculoskeletal, cardiovascular, and central nervous systems.

This project aims to explore the exercise habits and preferences of community-dwelling older adults with chronic pain. By identifying facilitating factors and barriers related to exercise, we can develop tailored exercise programs. These programs will promote healthier habits, allowing older adults to continue living independently in their communities and potentially delaying the need for long-term care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 or above
* Scored >6 in the Abbreviated Mental Test
* Can understand Cantonese
* Have a history of non-cancer pain in the past 6 months

Exclusion Criteria:

* Have a serious organic disease or malignant tumour
* Have a mental disorder diagnosed by neurologists or psychiatrists
* Have further medical/surgical treatment in two months or experienced drug addiction

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age: Participants are aged 60 years or above. Inclusion Criteria: Must score above 6 on the Abbreviated Mental Test, understand Cantonese, and have a history of non-cancer pain in the past 6 months.
  Exclusion Criteria: Excludes those with serious organic diseases, malignant tumors, diagnosed mental disorders, or recent drug addiction.
  Recruitment: Participants will be recruited from Neighborhood Elderly Centers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory | 1 year
  Participants, who are community-dwelling older adults with chronic pain, will be interviewed individually or in groups. During the 20-minute interviews, they will be asked about their pain situations, including pain intensity and sites of pain
Exercise habits and preferences | 1 year

IPD SHARING:
Plan to Share IPD: Undecided